CLINICAL TRIAL: NCT04224116
Title: Tranexamic Acid Contribution in the Prevention of Perioperative Bleeding in Pulmonary Resection Surgery
Brief Title: Tranexamic Acid Contribution in the Prevention of Perioperative Bleeding in Thoracic Surgery
Acronym: Bleeding
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, Amani Ben Haj Youssef, Tranexamic Acid Contribution in the Prevention of Perioperative Bleeding in Pulmonary Resection Surgery, University Tunis El Manar
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TA
Record Dates: First submitted 2019-10-01; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Bleeding
Keywords: tranexamic acid; Antifibrinolytic agents; bleeding; blood transfusion; thoracic surgery.
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: It's a randomized, double-blind, prospective study including patients over the age of 18 years old, programmed for potentially hemorrhagic thoracic surgery, such as pulmonary resection for aspergilloma, pulmonary tuberculosis, pleural decortication, lobectomy with parietectomy or redux. Demographic, clinical, biological data as well as transfusion requirements, blood loss and perioperative complications were identified.
  Two groups of patients:
  * TA group: receiving tranexamic acid (25mg/kg) in bolus at induction followed by 2mg/kg/h in continuous infusion until the end of the act.
  * Serum saline isotonic (SSI) group: placebo with isotonic saline serum.
Who Masked: Participant, Care Provider, Investigator
Masking Description: double blind investigation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group TA (Experimental): receiving tranexamic acid (25mg/kg) in bolus at induction followed by 2mg/kg/h in continuous infusion until the end of the act.
  Interventions: Drug: Tranexamic acid injection
- Group SSI (Placebo Comparator): Serum saline isotonic (SSI) group: placebo with isotonic saline serum.
  Interventions: Drug: SSI

INTERVENTIONS:
Drug: Tranexamic acid injection — to receive tranexamic acid (25mg/kg) in bolus at induction followed by 2mg/kg/h in continuous infusion until the end of the act.
  Other Names: EXACYL
  Arms: Group TA
Drug: SSI — Serum Salin isotonic injected
  Other Names: placebo
  Arms: Group SSI

SUMMARY:
Bleeding after thoracic surgery is a major cause of perioperative hemodynamic instability and transfusion requirement, which can lead to a rise of morbidity, mortality and costs.

The objective of this study is to evaluate the efficiency of tranexamic acid (TA) in the prevention of perioperative bleeding in thoracic hemorrhagic surgery.

DETAILED DESCRIPTION:
It's a randomized, double-blind, prospective study including patients over the age of 18 years old, programmed for potentially hemorrhagic thoracic surgery, such as pulmonary resection for aspergilloma, pulmonary tuberculosis, pleural decortication, lobectomy with parietectomy or redux. Demographic, clinical, biological data as well as transfusion requirements, blood loss and perioperative complications were identified.

Two groups of patients:

* TA group: receiving tranexamic acid (25mg/kg) in bolus at induction followed by 2mg/kg/h in continuous infusion until the end of the act.
* Serum saline isotonic (SSI) group: placebo with isotonic saline serum.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 18 years old, programmed for potentially hemorrhagic thoracic surgery, such as pulmonary resection for aspergilloma, pulmonary tuberculosis, pleural decortication, lobectomy with parietectomy or redux.

Exclusion Criteria:

* Patients who have had a major complication of surgery other than bleeding requiring revision within 24 hours or a complication related to anesthesia, and cases of non-compliance with the anesthetic protocol are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2019-10-02 (Actual); Study Completion 2019-10-02 (Actual)

PRIMARY OUTCOMES:
intraoperative bleeding volume | five hours
  The blood volume collected in the suction tanks and the operative drapes intraoperatively

SECONDARY OUTCOMES:
The number of red globular caps transfused for each group | one month
  transfusion if hemoglobin less than 7 g / dl
bleeding volume in the thoracic drains postoperatively | one month
  bleeding volume in the thoracic drains postoperatively every day

CONTACTS AND LOCATIONS:
Overall Officials: Tahar Mestiri, Professor, Principal Investigator — university Manar Tunis

IPD SHARING:
Plan to Share IPD: No